CLINICAL TRIAL: NCT05173272
Title: A Prospective Randomized Controlled Trials of Neoadjuvant Chemotherapy Combined With Serplulimab Followed by Concurrent Chemoradiation Versus Concurrent Chemoradiation Therapy Alone in Advanced Cervical Cancer
Brief Title: Induction Chemotherapy Combined With Immunotherapy Followed by Concurrent Chemoradiation in Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Guonan Zhang, Director, Head of Gynecologic Oncology Center, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2021-109
Record Dates: First submitted 2021-12-26; First posted 2021-12-29 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Neoadjuvant Therapy; Chemoradiotherapy; Brachytherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Neoadjuvant Therapy+CCRT (Experimental): Patients will be treated with 2 cycles of neoadjuvant chemotherapy (Cisplatin 50 mg/m^2 d1 q21+ Paclitaxel 175 mg/m^2 d1 q21) combined with serplulimab （300mg d1 q21）. After that, weekly cisplatin 30mg/m^2 for 4 or 5 weeks is administered concomitant with external beam radiotherapy (45-50.4Gy) in 1.8-2 daily fractions and a 10-20 Gy boost to reach a total dose of 65 Gy when there was unresectable lymph nodes. The primary cervical tumor is the boosted, using image guided 3D brachytherapy or 2D brachytherapy, with an additional 30-40 Gy to HRCTV (3D brachytherapy) or to point A (2D brachytherapy), to achieve a total dose of 80 Gy for small-volume cervical tumors or 85 Gy for larger-volume cervical tumors. All radiotherapy should be completed within eight weeks.
  Interventions: Drug: Neoadjuvant Therapy; Radiation: CCRT; Radiation: Brachytherapy
- Experimental: CCRT alone (Experimental): weekly cisplatin 40mg/m^2 for 4 or 5 weeks is administered concomitant with external beam radiotherapy (45-50.4Gy) in 1.8-2 daily fractions and a 10-20 Gy boost to reach a total dose of 65 Gy when there was unresectable lymph nodes. The primary cervical tumor is the boosted, using image guided 3D brachytherapy or 2D brachytherapy, with an additional 30-40 Gy to HRCTV (3D brachytherapy) or to point A (2D brachytherapy), to achieve a total dose of 80 Gy for small-volume cervical tumors or 85 Gy for larger-volume cervical tumors. All radiotherapy should be completed within eight weeks.
  Interventions: Radiation: CCRT; Radiation: Brachytherapy

INTERVENTIONS:
Drug: Neoadjuvant Therapy — Cisplatin 50 mg/m^2 d1 q21+ Paclitaxel 175 mg/m^2 d1 q21+serplulimab 300mg d1 q21
  Other Names: Neoadjuvant chemotherapy combined with Serplulimab
  Arms: Experimental: Neoadjuvant Therapy+CCRT
Radiation: CCRT — weekly cisplatin for 4 or 5 weeks is administered concomitant with EBRT (45-50.4Gy) in 1.8-2 daily fractions and a 10-20 Gy boost to reach a total dose of 65 Gy when there was unresectable lymph nodes.
  Other Names: chemoradiation
Radiation: Brachytherapy — The primary cervical tumor is the boosted, using image guided 3D brachytherapy or 2D brachytherapy, with an additional 30-40 Gy to HRCTV (3D brachytherapy) or to point A (2D brachytherapy), to achieve a total dose of 80 Gy for small-volume cervical tumors or 85 Gy for larger-volume cervical tumors.

SUMMARY:
The main objective of this study is to determine whether neoadjuvant chemotherapy combined with slulimumab sequential concurrent chemoradiotherapy versus concurrent chemoradiotherapy for locally advanced cervical cancer could improve progression-free survival rates.

Women in the experimental arm will receive neoadjuvant chemotherapy (cisplatin plus paclitaxel) combined with slulimumab every 21 days during 2 cycles followed by concurrent chemoradiation therapy. Women in the control arm will receive concurrent chemoradiation therapy alone.

286 patients will be recruited during 2 years, with 3 years of follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patients must have histologically confirmed cervical cancer with adenocarcinoma, adenosquamous or squamous histology and FIGO 2018 Ib3-IIIc2.
* According to the RECIST 1.1 standard, the subject must have at least one measurable target lesion
* No prior treatment
* Expected survival period ≥ 3 months
* ECOG score: 0-1
* No obvious signs of hematological diseases, ANC≥1.5×10^9/L, platelet count≥100×10^9/L, Hb≥90g/L, WBC≥3.0×10^9/L, and no bleeding tendency before enrollment;
* Adequate hepato-renal function is needed, including: Total bilirubin (TBIL)≤1.5×ULN (Gilbert syndrome allows ≤5×ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN Serum creatinine (Cr) ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50mL/min
* Cardiac Function: left ventricular ejection fraction (LVEF) >=50%;
* Patients voluntarily participated in the study and signed informed consent

Exclusion Criteria:

* Pregnant or breastfeeding female patients (women of child-bearing potential must confirm that the pregnancy test is negative within 7 days before the first administration. If it is positive, ultrasound examination must be performed to exclude pregnancy), or women of child-bearing potential who refused to receive contraceptive measures
* Combined with other malignant tumors, except for cured skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of any other part
* Existence of any bone marrow dysplasia and other abnormal hematopoietic diseases
* Active infections, HIV infections, and viral hepatitis that require systematic treatment
* Patients with≥Grade 1 peripheral neuropathy according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) Version 5.0
* Had severe cardiovascular diseases such as cerebrovascular accident, myocardial infarction, hypertension that cannot be controlled after drug intervention, unstable angina pectoris, heart failure (NYHA 2-4) and arrhythmia that need drug intervention within 6 months
* It is known to have a history of allergies to research drugs or drug components
* Has clinically significant thyroid dysfunction before enrollment;
* Has participated in other anti-tumor intervention clinical trials within 30 days before the first medication
* Have a clear history of dementia, mental state changes or any mental illness that will hinder understanding or informed consent
* The investigator believes that the patient is not suitable for participating in this clinical research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2027-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 36 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, or by histopathologic confirmation of suspected disease progression, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. Unequivocal progression of non-target lesions is also considered PD.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 48 months
  OS is the time from randomization to death due to any cause.
Objective Response Rate (ORR) | Up to approximately 36 months
  ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target and non-target lesions and also includes reduction of all nodal lesions to <10mm) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions and includes no unequivocal progression in non-target lesions) per RECIST 1.1.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 36 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guonan Zhang, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sicchuan cancer hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No